CLINICAL TRIAL: NCT07089108
Title: Validation of an Arabic Adaptation of the Naturalistic Observation Diagnostic Assessment (NODA) for Diagnosing Autism Spectrum Disorder in Saudi Arabia
Brief Title: Arabic NODA Validation Study for Autism Diagnosis in Saudi Arabia
Acronym: NODA-ARSA
Status: Completed | Type: Observational
Sponsor: Prince Sultan Military Medical City (Other)
Responsible Party: Principal Investigator, Fahad Alhusain, Research Scientist, Prince Sultan Military Medical City
Other Study IDs: PrinceSultanMilitaryMedCity
Record Dates: First submitted 2025-05-20; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-02

CONDITIONS: Autism Spectrum Disorder (ASD); Neurodevelopmental Disorders; Child Development Disorders, Pervasive
Keywords: Autism Spectrum Disorder; ASD; Autism Diagnosis; Telehealth; NODA; Naturalistic Observation Diagnostic Assessment; Arabic; Saudi Arabia; Cultural Adaptation; Remote Video Assessment; Early Childhood Development; Diagnostic Accuracy; Neurodevelopmental Disorders; Digital Health; Pediatric Autism
MeSH Terms: conditions — Autism Spectrum Disorder; Neurodevelopmental Disorders; Child Development Disorders, Pervasive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD Group: Children aged 6 months to 6 years with a confirmed diagnosis of Autism Spectrum Disorder (ASD) based on DSM-5 criteria and standardized tools (e.g., ADOS-2, ADI-R). Caregivers recorded four structured home videos using the Arabic NODA app to capture social communication and behavior for remote diagnostic evaluation.
  Interventions: Behavioral: Arabic NODA Video-Based Diagnostic Assessment
- Typically Developing Group: Children aged 6 months to 6 years with no known developmental, behavioral, or academic concerns and no family history of ASD. Participants were screened using the Arabic SCQ. Caregivers recorded four standardized home video scenarios using the Arabic NODA app for comparative assessment.
  Interventions: Behavioral: Arabic NODA Video-Based Diagnostic Assessment

INTERVENTIONS:
Behavioral: Arabic NODA Video-Based Diagnostic Assessment — NODA (Naturalistic Observation Diagnostic Assessment) is a telehealth-based diagnostic tool for Autism Spectrum Disorder (ASD) that guides caregivers to record structured home videos of their child's behavior using a smartphone app. In this study, a culturally adapted Arabic version of NODA was used to capture four standardized behavioral scenarios, which were later reviewed by licensed clinicians for diagnostic evaluation.
  Other Names: Naturalistic Observation Diagnostic Assessment; NODA

SUMMARY:
This study aims to validate the Arabic adaptation of the Naturalistic Observation Diagnostic Assessment (NODA), a telehealth tool designed to help diagnose Autism Spectrum Disorder (ASD) in young children. NODA guides parents to record home videos of their child in specific everyday situations, which are then reviewed remotely by trained clinicians. The study will compare the results from NODA video assessments to gold-standard in-person diagnostic evaluations. By testing the accuracy and feasibility of Arabic NODA in Saudi Arabia, this research may help improve access to early ASD diagnosis, especially for families in remote or underserved areas.

DETAILED DESCRIPTION:
This cross-sectional diagnostic validation study evaluates the Arabic adaptation of the Naturalistic Observation Diagnostic Assessment (NODA), a smartphone-based telehealth diagnostic tool for Autism Spectrum Disorder (ASD). The study employs a systematic cultural adaptation methodology including forward translation, expert panel review, back-translation, cognitive interviewing, and pilot testing to ensure cultural appropriateness for Saudi populations.

The validation phase involves 200 children (100 with confirmed ASD diagnoses, 100 typically developing controls, ages 6 months to 6 years) recruited from autism centers and pediatric clinics in Riyadh, Saudi Arabia. Caregivers use the Arabic NODA smartphone application to record four standardized behavioral scenarios in their home environment: family mealtime, play with others, play alone, and parent-reported concerns.

Two licensed clinicians, blinded to participant diagnostic status, independently review all video submissions through a secure web portal and provide diagnostic determinations based on DSM-5 criteria. Primary analysis compares NODA-based diagnoses to gold-standard clinical evaluations established through comprehensive in-person assessments using standardized tools (ADOS-2, ADI-R). Statistical analysis includes calculation of sensitivity, specificity, predictive values, inter-rater reliability, and receiver operating characteristic curves to establish diagnostic accuracy metrics and assess clinical utility for telehealth ASD diagnosis in Arabic-speaking populations.

ELIGIBILITY:
Inclusion Criteria:

* Age between 6 months and 6 years old
* For ASD group: Confirmed diagnosis of Autism Spectrum Disorder (ASD) based on DSM-5 criteria established through comprehensive clinical evaluation including standardized assessments (ADOS-2, ADI-R)
* For typically developing group: No developmental, behavioral, or academic concerns reported by parents or teachers; negative screening for ASD using Arabic Social Communication Questionnaire (SCQ)
* Parent or primary caregiver fluent in Arabic language
* Access to a smartphone with internet connectivity
* Ability to complete all four NODA video recording scenarios using the Arabic smartphone application

Exclusion Criteria:

* Significant visual or hearing impairments that would interfere with video-based behavioral assessment
* Major motor impairments that significantly limit the child's ability to interact socially or participate in video recording tasks
* Diagnosed genetic syndromes or neurological conditions unrelated to ASD
* Non-Arabic speaking household
* Inability to complete the required video recording protocol after training and support

Ages: 6 Months to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children aged 6 months to 6 years, including those with confirmed Autism Spectrum Disorder and typically developing controls. Participants are recruited from clinical autism centers, general pediatric clinics, and community settings in Riyadh, Saudi Arabia.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-08-21 (Actual); Study Completion 2022-12-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic Accuracy of Arabic NODA Compared to Gold-Standard ASD Diagnosis | Within 3 weeks of video submission
  This outcome will assess the diagnostic accuracy of the Arabic NODA system in identifying Autism Spectrum Disorder (ASD) in children aged 6 months to 6 years. Accuracy will be determined by comparing NODA-based diagnoses to gold-standard clinical diagnoses using DSM-5 criteria and standardized assessments (ADOS-2 and ADI-R). Metrics will include sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and overall percent agreement.

SECONDARY OUTCOMES:
Inter-rater Reliability Between Independent NODA Clinicians | Within 3 weeks of video submission
  Two licensed clinicians will independently review the NODA videos and provide ASD diagnostic determinations. The inter-rater reliability will be evaluated using percent agreement and Cohen's kappa coefficient. Intraclass correlation coefficients (ICC) may be calculated for DSM-5 domain scores across reviewers.
Video Completion Rate | Within 3 weeks of enrollment
  Proportion of families who successfully complete all four Arabic NODA video scenarios using the smartphone application. This feasibility metric will be calculated as the percentage of enrolled families who submit all required video recordings within the specified timeframe.
Time to Video Completion | Within 3 weeks of enrollment
  Duration from study enrollment to successful submission of all four required video scenarios. This will be measured in days and reported as mean, median, and range to assess the practical timeline for completing the Arabic NODA assessment process.
Technical Difficulties Frequency | Within 3 weeks of enrollment
  Number and type of technical challenges encountered during the video recording process. This will include frequency of app-related issues, video quality problems, upload failures, and user support requests. Data will be categorized by difficulty type and severity.
Parent Satisfaction with the Arabic NODA Application | Within 1 week after video submission is completed
  Parents will complete a satisfaction survey using a 5-point Likert scale (1 = very dissatisfied, 5 = very satisfied) after submitting NODA videos. The survey will assess usability, clarity of instructions, cultural appropriateness, and overall satisfaction with the video-guided diagnostic process. Higher scores indicate better satisfaction.
Clinician Confidence in Diagnostic Decision Based on Arabic NODA Videos | Within 1 week after clinician video review completion
  After reviewing each child's videos, clinicians will rate their confidence in their diagnostic decision on a 5-point scale (1 = extremely low confidence, 5 = extremely high confidence). This outcome evaluates the clinical utility and perceived sufficiency of information provided by the Arabic NODA system. Higher scores indicate greater clinician confidence.

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Sultan Military Medical City, Riyadh, Riyadh Region, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to the sensitive nature of the data, which includes video recordings of young children in home environments. These materials are difficult to fully de-identify and are subject to strict ethical and privacy protections under local regulations and IRB oversight.